CLINICAL TRIAL: NCT03609320
Title: Improving HPV Vaccination Delivery in Pediatric Primary Care: The STOP-HPV Trial 5. Single Arm Evaluation of the Bundle (Communication Skills, Performance Feedback and Prompts)
Brief Title: The STOP-HPV Trial 5: Single Arm Evaluation of the Bundle
Acronym: STOP_HPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Academy of Pediatrics (Other); University of Pennsylvania (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, Executive Vice-Chair and Vice-Chair for Research, Department of Pediatrics, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01CA202261 (NIH); R01CA202261 (NIH)
Record Dates: First submitted 2018-06-29; First posted 2018-08-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Immunization; Vaccination
Keywords: HPV; Vaccination; Practice Based Intervention

STUDY DESIGN:
Intervention Model Description: This single-arm study embedded within a 2-arm cluster RCT will test the difference in the rate of missed opportunities pre- and post-implementation of a 3-component intervention including communication skills, performance feedback, and prompts. These three interventions will be implemented together in practices that previously received standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): These practices, which previously received standard of care, will receive The STOP-HPV Trial 5: Bundle Intervention
  Interventions: Behavioral: The STOP-HPV Trial 5: Bundle Intervention

INTERVENTIONS:
Behavioral: The STOP-HPV Trial 5: Bundle Intervention — This intervention will implement a 3-component bundle intervention (communication skills training, performance feedback and prompts) together in practices that previously received standard of care.

SUMMARY:
Most adolescents who receive human papillomavirus (HPV) vaccine are vaccinated in pediatric practices, yet missed opportunities (MOs) for HPV vaccination occur often and lead to low HPV vaccination rates. This single-arm study (embedded within arm 2 of a 2-arm cluster randomized clinical trial (RCT)) will test the effectiveness (and cost-effectiveness) of a bundled intervention (HPV vaccine communication, performance feedback reports and provider prompts), in practices that previously received standard of care, to reduce MOs and increase HPV vaccination rates.

DETAILED DESCRIPTION:
HPV vaccine rates remain lower than rates for other adolescent vaccines. Missed opportunities (MOs) are healthcare visits during which a patient is eligible, but does not receive a vaccine. MOs for vaccination contribute strongly to low HPV vaccination rates. This single-arm study (embedded within arm 2 of a 2-arm cluster RCT) will implement a 3-component bundle intervention together in practices that previously received standard of care. This study will test the effectiveness (and cost-effectiveness) of the bundled intervention, which trains providers in HPV vaccine communication (done through online educational modules and live office practice sessions), provides performance feedback reports (that pull from electronic health record (EHR) data, and compare participants' performance to their own previous performance and performance of others) and provider prompts (via EHR and also office staff prompts, e.g., placing Vaccine Information Statements (VISs) on desk) to reduce MOs and increase HPV vaccination rates. Throughout the intervention participants will also receive weekly text message mini-lessons that will remind participants of the project.

ELIGIBILITY:
Practice Inclusion Criteria:

* The practice provides HPV vaccination services to adolescents.
* The practice is part of Physician's Computer Company (PCC), Office Practicum (OP) or (a) yet-to-be selected health system(s).
* The practice has had the same EHR system in place for a year or more (with special consideration on a case by case basis if they are close to but not do not reach a year).
* The practice agrees to not participate in other HPV-related QI projects or research interventions during the study period (with special consideration on a case by case basis).

Practice Exclusion Criteria:

* The practice plans to change EHR systems in the next three years.
* The practice participated in the last year, is currently engaged in, or plans to participate in an office-based HPV-related quality improvement (QI) project or research intervention during the study period (with special consideration on a case by case basis).
* Estimated 20% or more of adolescents at the practice receive HPV vaccinations at schools or health department clinics (given standard practice and published data, the investigators expect that few to no practices will need to be excluded based on this restriction).

Patient inclusion criteria:

-All patients of participating practices (intervention and comparison) aged 11-17 years who have at least 1 visit to the practice within the past two years.

Patient exclusion criteria:

-None apart from age of patients (above).

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-08-09 (Estimated); Study Completion 2022-08-09 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of missed vaccination opportunities among all clinicians | The 12-month period immediately preceding initiation of the bundle and the 6-month bundle period, excluding the 6-week ramp-up
  Change in the rate of missed vaccination opportunities from the 6 month bundle intervention period versus the 12 month period preceding the bundle period among all clinicians.
Change in the rate of missed vaccination opportunities among consenting clinicians | The 12-month period immediately preceding initiation of the bundle and the 6-month bundle period, excluding the 6-week ramp-up
  Change in the rate of missed vaccination opportunities from the 6 month bundle intervention period versus the 12 month period preceding the bundle period among consenting clinicians.

SECONDARY OUTCOMES:
Change in the rate of missed vaccination opportunities among all clinicians. | From months 0 (baseline) through month 28 of study activities. Study activities were paused for a 15 month period during the pandemic.
  Change in the rate of missed vaccination opportunities among all clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- American Academy of Pediatrics, Itasca, Illinois, United States

IPD SHARING:
Plan to Share IPD: No